CLINICAL TRIAL: NCT00286039
Title: Plasma Citrulline Level in Relation to Absorptive Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2005/163
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Intestinal Failure
MeSH Terms: conditions — Intestinal Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling is used.

SUMMARY:
Correlation between determination of citrulline in plasma or dried blood

Reference ranges for healthy children and babies

Longitudinal follow-up of citrulline in preterm babies

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years
* preterm babies up to 1.500g
* preterm babies over 1.500g

Exclusion Criteria:

* gastro-intestinal problems (except for the preterm babies)
* congenital metabolic disorders
* dysfunction of the liver or kidneys
* congenital defects

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2005-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Correlation between determination of citrulline in plasma or dried blood | Untill end of study
Reference ranges for healthy children and babies | Until end of study
Longitudinal follow-up of citrulline in preterm babies | Untill end of study

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Robberecht, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be